CLINICAL TRIAL: NCT02782936
Title: Impact of Gas Masks on Index of Efforts and Breathing Pattern
Brief Title: The Gas Mask: the Effects on Respiration!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Pierre-Alexandre Bouchard, RT. (Unknown); Captain (Ret) Stephane Bourassa, RN. (Unknown)
Responsible Party: Principal Investigator, François Lellouche, Physician, Laval University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 21140; 2015-2448 (Other: CRIUCPQ)
Record Dates: First submitted 2016-05-19; First posted 2016-05-26 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Work of Breathing
Keywords: Work of Breathing; Hypoxemia; Respiratory Acidosis; Respiratory effort
MeSH Terms: conditions — Hypoxia; Acidosis, Respiratory | interventions — Respiratory Protective Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Baseline (Experimental): Randomised baseline without and with gas mask.
  Interventions: Other: measurement of the work of breathing; Device: Gas mask
- Induced Hypoxemia (Experimental): Randomised hypoxemia: i. without gas mask; ii. with gas mask; and iii. correction with FreeO2 and gas mask.
  Interventions: Other: measurement of the work of breathing; Device: Gas mask
- Effort (Experimental): Randomised effort without and with gas mask
  Interventions: Other: measurement of the work of breathing; Device: Gas mask

INTERVENTIONS:
Other: measurement of the work of breathing — We have been evaluating breathing patterns, index of respiratory efforts and blood gases in all randomized conditions. A gas mask has been used mask (C4, Airboss Defence, Bromont, Canada).
  Airway pressure, inspiratory and expiratory flows have been measured. An esophageal catheter has been introduced at the beginning of the study to measure esophageal pressure (Peso) and calculate indexes of respiratory effort (PTPeso, WOB). SpO2 has been continuously measured and capillary blood bases were drawn at the end of each condition. Each condition lasted 10 minutes, data of the last 2 minutes at a steady state has been considered for analyses.
Device: Gas mask — During the conditions that involved a gas mask, the measurement of the work of breathing is achieved with a oesophageal catheter and two disposable pneumotachs. While the oesophageal catheter has been fixed to the mandibular with an hypo-allergic tape, the two pneumotachs are hooked respectively on the canister and exhalation port of the gas mask. Investigators have induced the hypoxemia with a mixture nitreous and medical gas in a plastic bag that has been setted up to the canister. The FiO2 level has been kept to 14 percent.
  Other Names: Canadian Gas Mask C-4 manufactured by Airboss Defence, Bromont, Québec, Canada.

SUMMARY:
Background: The gas mask is used to protect military and non-military subjects exposed to respiratory hazards (CBRN agents). The aim of the study was to evaluate the impact of the gas mask on respiratory patterns and indexes of the respiratory effort. Methods: We are completing our study with 14 healthy subjects to evaluate breathing patterns, index of respiratory efforts and blood gases. Seven conditions have been tested in a randomized order: at rest, during effort (on a tread mill, standardized at 7 METs for all subjects) and during induced hypoxemia with and without a mask (C4, Airboss Defence, Bromont, Canada). Airway pressure, inspiratory and expiratory flows were measured. An esophageal catheter was introduced at the beginning of the study to measure esophageal pressure (Peso) and calculate indexes of respiratory effort (PTPeso, WOB). SpO2 was continuously measured and capillary blood bases were drawn at the end of each condition. Each condition lasted 10 minutes, data of the last 2 minutes at a steady state were considered for analyses. Results: The preliminary analyses based on 10 subjects are presented here. Comparing the wearing of the gas mask and without, most of the respiratory index increased in the tested conditions (at rest, during induced hypoxemia and during effort). At rest, in 8 out of 10 healthy subject the indexes of effort were higher with the gas mask, a statistical trend was observed with the WOB (0.22±0.13 vs. 0.28±0.10 J/cycle; p = 0.059), the PTPes (101±35 vs. 122±47 cmH2O*s; p=0.21) and SwingPeso (4.4±2.0 vs. 5.3±2.0 cmH2O; p=0.13). During the effort, the respiratory index increased (WOB 4.0±2.6 vs. 5.6±3.2; p=0.10; PTPeso 406±211 vs. 606±65; p=0.04; SwingPeso 14.8±8.1 vs. 21.8±9.0; p=0.13). There was no difference for the breathing pattern and arterial blood gases data with and without mask. Data for induced hypoxemia are under analysis. We measured on bench the inspiratory and expiratory resistances of the tested gas mask (C4: inspiratory resistances = 3.2 cmH2O at 1 L/sec; expiratory resistances = 0.9 cmH2O at 1 L/sec). This may explain in part the increased work of breathing with masks. Conclusions: This study demonstrated an increase of the indexes of respiratory effort during an exercise with the gas mask. This study is the first to directly assess the indexes of efforts with esophageal pressure in this situation. Our results and method may be used as a reference for evaluating tolerance with different designs of gas masks.

DETAILED DESCRIPTION:
The principal way of penetration of CBRNE agents is the respiratory system. The current technology of a gas mask has been used to protect the respiratory system as far back as the First World War. That originated from Dr Cluny Macpherson's initiatives whom was a Canadian military physician.

The military gas mask is part of the respirator classification but owes its specific features. Conventionally, the military gas mask covers a large spectrum of protection aspects and matched with their specific canisters. Consequently, gas masks are usually studied separately from other respirators and Self-Contained Breathing Apparatus (SBCA).

The gas mask design and its components may lead to these respiratory load issues. At rest and effort, what would be the impacts for the work of breathing and gas exchange? In order to avoid hypoxemia and hyperoxia, what would be the optimal means to restore proper oxygenation? We hypothesised: i. on a heightened WOB and the respiratory demands related to wear of the gas mask; ii. An occurrence of hypoxemia will be manifesting during a continuous period at both at rest and effort.

Our goal was to measure the impact of the work of breathing and the gas exchange for a gas mask user. We also measured what was the optimal means for correcting the hypoxemia with a subject.

14 Male Human Subjects participated in a comparison and single-blind randomized experimental study. That was approved by the Ethical Review Committee. All male subjects were in averaged age of 38.9±5 year old and a FEV1 4.60±0.70 Liter. A written consent was obtained for all the subjects prior their acceptance. No rejection happened during the recruiting. The eligibility criteria were: i. No significant cardiac and respiratory diseases known; ii. No epilepsy background; iii. No severe pathology requiring medication; iv. No pregnancy for woman; v. Face medium - size in relation of the gas mask. The exclusion criteria were: i. Refusals relate to wear the oesophageal catheter and for capillary punctures; ii. Claustrophobia; iii. Oesophageal wounds backgrounds; iv. No coronary background and stroke history; v. No face morphology incompatibility with the mask. Spirometry and usual health screening was also done before starting the clinical trial.

Design comprised seven 10-minute testing conditions split in two parts. Five were at rest and sitting on a chair: i. Baseline without gas mask; ii. Baseline with gas mask; iii. Hypoxemia without mask; iv. Hypoxemia with gas mask; and v. Hypoxemia corrected. Two effort conditions were programmed at 7 METS Effort Zone and were performed on Treadmill (Constant 3 MPH speed and 10% inclination). These were with and without the gas mask. Between the rest-condition a 5-minute wash-out took place while for the effort a ten-minute was applied.

Three five-minute periods was followed to record blood pressure and pulse during the conditions. SpO2 was continuously measured with Free O2 during condition while the Massimo was employed also at the beginning both the inclusion and at the each three hypoxemia condition (Radical - Signal Extraction Pulse Oximeter). During effort, they were taken at each two-minute, starting at a zero starting point. Capillary punctures were done at the end of each condition.

Our main measurements were the WOB performed with a continuous recording of Peso pressure and respiratory volumes. Software Acknowledge, version 3.9 served as acquisition data system and analysis were achieved with a 4.2 version and a free-trial WOB calculus system, named RESPMAT. That was obtained from Maynaud and al. [2]. As power source, we used a BIOPAC (MP100, Santa Barbara, Californie, USA, 200 Hertz), four differential sensors (Validyne : 1x MP45±100 cmH2O; 2x MP??±5 cmH2O; 1x MP100±100 cmH2O) and four Carrier D-Modulators (Validyne, CT-15,120 Volt, 60 Hertz, 5Watts, Model CD15-A-2-A-1).

Single esophageal catheter (Type Cooper, French caliber #5) and disposable pneumotachs were used. Lidocain spray and K-Y gel were applied during the insertion of the catheter. Its placement was done at 37.6±5.7 cm across the subject and a Mueller test was performed for each subject. In regard of spontaneous breathing, an Hudson mask was used while a C-4 Gas Mask with a canister was employed (Manufacturer: Airboss Defence, Bromont, Canada). Hypoxemia mixture was home-design with usual nitrous and medical gas and maintaining a FiO2 target at 14%. Prototyped Free O2 System was employed for the correction of the hypoxemia.

ELIGIBILITY:
Inclusion

* Having no significant cardiac and respiratory pathology
* Having no history of epilepsy
* Having no severe and chronic pathology that requires medication
* Not being pregnant
* Face size: medium

Exclusion

* Refuse to participate in the study for one of the following reasons: i. wearing a oesophageal catheter; ii. wearing the gas mask; iii. giving blood sample; iv. claustrophobia.
* Oesophageal background wounds
* Facial anthropometrical issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
indexes of respiratory effort | 10 minutes
  In this study, we speculate the work of breathing is increasing with the use of a gas mask at rest, under hypoxemia condition and during physical effort.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Lellouche, Doctorate, Principal Investigator — Institut de Recherche Universitaire de Cardiologie et Pneumologie de Québec
Locations (1):
- Institut de recheche universitaire de cardiologie et pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bourassa S, Bouchard PA, Dauphin M, Lellouche F. Oxygen Conservation Methods With Automated Titration. Respir Care. 2020 Oct;65(10):1433-1442. doi: 10.4187/respcare.07240. Epub 2020 Feb 18. PMID 32071135
- [Derived] Bourassa S, Bouchard PA, Lellouche F. Impact of Gas Masks on Work of Breathing, Breathing Patterns, and Gas Exchange in Healthy Subjects. Respir Care. 2018 Nov;63(11):1350-1359. doi: 10.4187/respcare.06027. Epub 2018 Jul 31. PMID 30065082